CLINICAL TRIAL: NCT02755987
Title: Expanded Access to ANG1005 for an Individual Patient With Recurrent WHO Grade III Anaplastic Astrocytoma; Expanded Access to ANG1005 for an Individual Patient With Recurrent WHO Grade III Anaplastic Oligodendroglioma; Expanded Access to ANG1005 for an Individual Breast Cancer Patient With Recurrent Brain Metastases and Leptomeningeal Carcinomatosis.
Brief Title: Expanded Access to ANG1005 for Individual Patients
Status: No longer available | Type: Expanded Access
Sponsor: Angiochem Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ANG1005-EAP-01, EAP-02, EAP-03
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Breast Cancer With Recurrent Brain Metastases; Leptomeningeal Carcinomatosis
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Meningeal Carcinomatosis | interventions — paclitaxel-Angiopep-2 conjugate

INTERVENTIONS:
Drug: ANG1005

SUMMARY:
This is an expanded access study with ANG1005 treatment for two individual patients from Protocol ANG1005-CLN-03 with WHO Grade III Anaplastic Astrocytoma and WHO Grade III Anaplastic Oligodendroglioma and one individual patient from Protocol ANG1005-CLN-04 with Recurrent Brain Metastases and Leptomeningeal Carcinomatosis.

ELIGIBILITY:
Inclusion Criteria:

1. Neurologically stable
2. Karnofsky performance status (KPS) ≥ 80
3. Adequate laboratory results

Exclusion Criteria:

1. Radiotherapy within 3 months.
2. Evidence of significant intracranial hemorrhage
3. NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0 Grade ≥ 2 neuropathy
4. Inadequate bone marrow reserve
5. Any evidence of severe or uncontrolled disease

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UC Irvine Health, Orange, California
  - Univeristy of Texas Health Science Center in San Antonio, San Antonio, Texas